CLINICAL TRIAL: NCT06813729
Title: Effects of Shotblocker® and Manual Pressure on Pain During the Administration of Vaccine in Infants
Brief Title: Effects of Shotblocker® and Manual Pressure on Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Nihal Taskiran, Aydin Adnan Menderes University, Aydin Adnan Menderes University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: E-79593712-605.99
Record Dates: First submitted 2025-01-29; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Healthy Volunteers; Infant; Vaccine; Pain
Keywords: pain; vaccine; shotblocker; manuel pressure; infant
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Trial
Who Masked: Participant
Masking Description: Infants who met the inclusion criteria and were scheduled for the PCV vaccine injection were assigned to one of three groups: Shotblocker®, manual pressure, or a control group (which received the standard injection technique). To address gender differences, infants were first categorized by gender and then randomly assigned to the three groups using block randomization. To ensure fairness and minimize bias, labels for each group (Shotblocker®, manual pressure, and control) were written on papers of the same color and shape, placed into separate pink and blue boxes. During the vaccination process, the group assignment was determined by a lottery that the mother drew from just before the procedure. Mothers of girls were instructed to draw from the pink box, while mothers of boys drew from the blue box. Each group consisted of 34 infants, with an equal distribution of 17 females and 17 males.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- The Shotblocker® Group (Experimental): Shotblocker® is a small, flexible plastic device designed to be drug-free, featuring multiple rounded points on the bottom that come into contact with the skin. It also has a central hole for injection administration.
  Interventions: Biological: Shotblocker
- The Manuel Pressure Group (Experimental): nurse held the infants' leg for the injection, 10-second manual pressure was applied on the vaccine injection site by the experienced nurse before pneumococcal conjugate vaccine
  Interventions: Biological: Manuel Pressure
- The Control Group (No Intervention): The infant was first placed on the examination table. To calm the infant, the mother was asked to hold the infants' hands and talk to him/her. Distraction method was not employed for the infants in this group, and while one nurse held the infants' leg for the injection, the experienced nurse administered the pneumococcal conjugate vaccine (0.5 ml, IM, Vastus Lateralis Site).

INTERVENTIONS:
Biological: Shotblocker — The infant was first placed on the examination table. To calm the infant, the mother was asked to hold the infants' hands and talk to him/her. Before the injection, while one nurse held the infants' leg for the injection, Shotblocker® was applied to the skin by the experienced nurse ensuring that the points were in direct contact. Then, the nurse administered the pneumococcal conjugate vaccine (0.5 ml, IM, Vastus Lateralis Site) through the central hole. After each use, the Shotblocker® was disinfected with 70% alcohol before being used on another infant.
  Arms: The Shotblocker® Group
Biological: Manuel Pressure — The infant was first placed on the examination table. To calm the infant, the mother was asked to hold the infants' hands and talk to him/her. Next, while one nurse held the infants' leg for the injection, 10-second manual pressure was applied on the vaccine injection site by the experienced nurse. Then pneumococcal conjugate vaccine was administered in accordance with the standard injection technique (0.5 ml, IM, Vastus Lateralis Site).
  Arms: The Manuel Pressure Group

SUMMARY:
Aim This randomized controlled experimental study was conducted to determine the effect of ShotBlocker® and manual pressure application on pain in the application of Conjugated Pneumococcal Vaccine (PCV).

The following hypotheses were determined for the study; Hypothesis 1: Pain scores of infants are lower in the manual pressure group than in the control group during the administration of PCV.

Hypothesis 2: Pain scores of infants are lower in Shotblocker® group than in the control group during the administration of PCV.

Hypothesis 3: Manual pressure is more effective than Shotblocker® in infants to reducing pain during the administration of PCV.

DETAILED DESCRIPTION:
The study was carried out at three family health centers, all with the same nurse administering care. Infant who were 4 months old and scheduled to receive the PCV vaccine were eligible for participation. The data were collected using a questionnaire form and the Neonatal Infant Pain Scale (NIPS).

A standard procedure was followed for all infants, which included bringing the infant and mothers into the vaccination room, providing information about the vaccine, introducing the researcher, and obtaining informed consent. Infants were assigned to groups based on randomization. To control factors related to the application process (such as injection technique and communication approach), vaccines were administered by same experienced nurse working at the family center where the research was conducted.

A video camera with a 5X optical zoom support (Samsung M51 brand smartphone) was used to record vaccine injections. It was placed on a tripod across the stretcher where the infants were vaccinated. Each infant was recorded for during vaccination, and 2 min after vaccination.

Written approval was obtained from the Ethics Committee (2021/279) and institution where the study was conducted (E-79593712-605.99). The nurse researcher informed infants' mothers about the study. Upon agreement from mothers, written consent forms were obtained.

Data were analyzed using SPSS for Windows version 25.0 (IBM, Armonk, NY). Numeric variables are presented as counts, percentages, means, standard deviations, and min-max values. The assumption of normal distribution was checked with the Shapiro-Wilk test, and the assumption of homogeneity of variances was controlled with the Levene test. To compare pain scores after vaccination, a paired sample t-test was used. In cases where the data showed a normal distribution and there were more than two independent groups, a one-way analysis of variance (ANOVA) test was employed. A significance level of p < .05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Infant who were 4 months old
* who receive the pneumococcal conjugate vaccine receive
* healthly infant, free from systemic illnesses
* accompanied by their mothers
* attending the center for routine vaccination

Exclusion Criteria:

* who have serious congenital malformations
* who have neurodevelopmental delays
* who have serious congenital malformations
* who have febrile conditions
* who have a history of circulatory or peripheral vascular issues
* who had taken sedatives, hypnotics, or systemic pain relievers within the last 6 hours
* infant who cried before receiving the vaccine

Ages: 4 Months to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Pain mean score | immediately after the pneumococcal conjugate vaccination
  The Neonatal Infant Pain Scale total mean score of infants are lower in the manual pressure and shotbocker groups than in the control group during the administration of PCV.

CONTACTS AND LOCATIONS:
Locations (1):
- Soma Family Health Center No. 3, Manisa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kislali Tas S, Sari D, Taskiran N. Reducing Vaccination Pain in Infants: A Randomized Controlled Trial on the Effects of ShotBlocker and Manual Pressure. Clin Pediatr (Phila). 2025 Oct 29:99228251387875. doi: 10.1177/00099228251387875. Online ahead of print. PMID 41159533